## **Exercise as Medicine: A Non-Pharmacological Approach to Menopausal Symptoms**

Date: 01-11-2025

## Data analysis and statistics

Statistics will be computed using IBM SPSS Statistics (New York, USA). Pre- and post-intervention results will be analysed using the Wilcoxon signed-rank test. To determine if there are statistically significant differences between the groups, the Kruskal-Wallis test (H-test) will be used. Due to the explorative nature of the study and cohort design no sample size calculation will be performed.